CLINICAL TRIAL: NCT03935607
Title: The Pseudo-Oligohydramnios/Hidden Pocket Study: The Added Contribution of Transvaginal Sonographic Evaluation of Amniotic Fluid Index
Brief Title: The Added Contribution of Transvaginal Sonographic Evaluation of Amniotic Fluid Index
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal Investigator, Rambam Health Care Campus
Other Study IDs: 0017-19-RMB
Record Dates: First submitted 2019-04-25; First posted 2019-05-02 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Oligohydramnios
MeSH Terms: conditions — Oligohydramnios

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal amniotic fluid index: Patients with an amniotic fluid index of between 5-24 centimeters according to transabdominal sonography.
  Interventions: Diagnostic Test: Transvaginal sonography
- Oligohydramnios: Patients with an amniotic fluid index of lss than 5 centimeters according to transabdominal sonography.
  Interventions: Diagnostic Test: Transvaginal sonography

INTERVENTIONS:
Diagnostic Test: Transvaginal sonography — Transvaginal sonography for the evaluation of an amniotic fluid pocket preceding the fetal presenting part.

SUMMARY:
The current study is based on the use of transvaginal sonography in the evaluation of oligohydramnios. Patients will be recruited after amniotic fluid index evaluation according to transabdominal sonography. After obtaining informed consent, transvaginal sonography will be used to evaluate and measure a possible amniotic fluid pocket that may precede the fetal presenting part.

DETAILED DESCRIPTION:
Background Normal amniotic fluid volume varies across gestation (Ounpraseuth 2017). Abnormal amniotic fluid volume has been associated with a variety of adverse pregnancy outcomes (Shrem 2016). In clinical practice, the amniotic fluid volume is a component of the biophysical profile which provides information on fetal well-being.

Transabdominal ultrasound is used to assess quantitatively the amniotic fluid volume, most commonly by either the Amniotic Fluid Index (AFI) or the Maximum Vertical Pocket (MVP) methods.

The value of the AFI method has been questioned in several studies, which have shown that an abnormal test, low or high, is neither highly accurate nor predictive of adverse outcome. Many pregnancies with normal AFI will be falsely characterized as abnormal, and a large number with truly abnormal AFI will be missed (Magann 1994, Chauhan 1997).

The MVP measurement may be preferred over the AFI method. A 2008 systematic review of randomized trials found that use of the AFI increased the rate of diagnosis of oligohydramnios (RR 2.3), induction of labor (RR 2.1), and cesarean delivery for fetal distress (RR 1.5) (Nabhan 2008).

Rationale and Hypothesis of the Study Recently, our group observed that when transvaginal ultrasound is being performed to non-laboring pregnant women at term for other obstetrical indications, there is a large amniotic fluid pocket above the internal cervical os and below the fetal presenting part. Due to the unique location of this pocket, we hypothesized that transvaginal ultrasound may provide better information than transabdominal ultrasound on amniotic fluid volume, particularly in cases when suspecting abnormal low amniotic fluid volume.

Data Collection

1. Maternal and fetal characteristics Data related to the fetomaternal antenatal, intrapartum and postpartum course will be recorded prospectively.
2. Ultrasound assessment Each eligible woman in the study population group will be asked to undergo prenatal ultrasound examination twice. The first ultrasound examination is a routine transabdominal ultrasound examination that is carried out to assess fetal growth and well-being. This is to be continued with a second transvaginal ultrasound, with a specific focus on the amniotic fluid pocket, that is; the distance in centimetres between the fetal presenting part and the internal cervical os. The second transvaginal ultrasound will be performed for the purpose of the study only, and by one other research team member that is blinded to the first routine transabdominal ultrasound. The entire length of the study, combining the transabdominal and transvaginal ultrasounds, is expected to take on the average around 15 min.

Ultrasound Equipment and Safety Considerations In their 2011 statement, The International Society of Ultrasound in Obstetrics and Gynaecology (ISUOG) and World Federation of Ultrasound in Medicine and Biology (WFUMB) consider ultrasonography to be safe for use during clinical practice (ISUOG 2011).

Statistical analyses and sample size For sample size calculation, and given a 20% rate of induction of labor, of which 3% are due to abnormal low amniotic fluid volume (oligohydramnios), a sample size of 1000 women is required.

Feasibility of the Study Considering the high volume of maternal care here at Rambam Health Care Campus, and that every year there are around 5,000 births and nearly double routine cares, the recruitment process for the current study is feasible.

Expected Duration of the Study The recruitment for the study is expected to take place over 12 months with an additional 3-6 months after recruitment for data analysis before publication.

Funding Women will be recruited while approaching Rambam Health Care Campus for their routine obstetric care. Ultrasound examinations will be carried out using existing operational ultrasound equipments within the obstetric department at Rambam Health Care Campus. For both, the recruitment and the ultrasound examinations, no extra funding is currently required.

Public Health Interest Identifying new ultrasound variables that can assist in quantifying amniotic fluid volume, as the one suggested in the current study, is of great importance and may provide invaluable information into the overall future care and decision-making around the time of delivery, especially whether or not to induce labor in women with suspected oligohydramnios. Thus, it may assist in creating future recommendations for pregnant women and improved healthcare standards during the delivery process.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at term beyond 37 weeks' gestation
* Presented to our hospital for their routine care or prior to induction of labor
* Singleton pregnancy
* Planned for vaginal delivery
* Non-laboring women with non-engaged fetal presenting part

Exclusion Criteria:

* Pregnant women under 37 weeks' gestation
* Planned cesarean deliveries
* Laboring women with engaged fetal presenting part
* Multiple gestation

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Prgenancy
Study Population: Women who meet the above inclusion criteria will be asked to participate in the study and to provide a written informed consent. This study, under no circumstances, will alter the participants routine care.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Amniotic Fluid Fore-Pocket | Up to 30 minutes from the beginning of patient evaluation.
  Measurement of amniotic fluid pocket preceding fetal presenting part.

SECONDARY OUTCOMES:
Mode of delivery | From time of induction up to 48 hours postpartum
  Vaginal delivery, vacuum assisted delivery, cesarean section.
pH level | From the time of delivery up to 30 days postpartum
  Umbilical artery pH level
1 minute Apgar score | From the time of delivery up to 30 days postpartum
  Neonatal 1st minute Apgar score
5 minute Apgar score | From the time of delivery up to 30 days postpartum
  Neonatal 5th minute Apgar score
Neonatal intensive care unit admission | From the time of delivery up to 30 days postpartum
  Rate of neonatal intensive care unit admission

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided